CLINICAL TRIAL: NCT04387435
Title: A Feasibility Study to Evaluate the Safety and Effect of the Optimization of Vagus Nerve Stimulation in Epileptic Patients to Induce Cardioprotection
Brief Title: Optimization of VNS in Epileptic Patients to Induce Cardioprotection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olujimi Ajijola, MD, PhD, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-002279; OT2OD028201 (NIH)
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy; Sudden Cardiac Death
Keywords: Vagus Nerve Stimulation (VNS); Neuromodulation; Autonomics
MeSH Terms: conditions — Epilepsy; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): Single arm
  Interventions: Other: A change or titration in the current or frequency settings of the VNS therapy system.

INTERVENTIONS:
Other: A change or titration in the current or frequency settings of the VNS therapy system. — The study treatment involves changing the output current or frequency of the default device settings in a FDA approved device for VNS therapy. The proposed frequency changes in this study are within the FDA approved output current and frequency levels.

SUMMARY:
This study is a non-randomized, prospective study in patients with a diagnosis of epilepsy and previously implanted FDA approved Vagus Nerve Stimulation (VNS) devices. The goal of this clinical investigation is to evaluate the effects of adjusting vagus nerve stimulation parameters to engage cardioprotective effects.

DETAILED DESCRIPTION:
Epilepsy patients are at increased risk for sudden cardiac death. Mechanisms behind this predisposition is poorly understood but parasympathetic dysfunction is heavily implicated. Vagus Nerve Stimulation (VNS) protocols currently set for seizure management are poorly optimized for cardioprotection, therefore this patient population presents a unique opportunity to assess VNS control of cardiac function, when VNS is appropriately titrated for cardiac and seizure benefit.

This study will enroll 12 patients with a diagnosis of epilepsy and previously implanted FDA approved VNS devices. The study will last up to 9 weeks and the patient will undergo changes to their VNS settings during autonomic testing and cardiopulmonary testing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of refractory epilepsy and implanted with a VNS device or are scheduled to be implanted with a VNS device.
* 18 years of age or older
* Subjects must demonstrate willingness and ability to comply with study requirements

Exclusion Criteria:

* Other implantable neuromodulatory device (e.g., brain stimulator)
* Treatment with cholinergic or anticholinergic medication in the past month
* Pre-existing cardiac arrhythmia or presence of cardiac pacemaker/defibrillator
* History of dysautonomias
* History of vasovagal syncope
* Progressive neurological diseases other than epilepsy
* Women that are pregnant
* Cognitive or psychiatric deficit that in the investigator's judgment would interfere with the subject's ability to accurately complete study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olujimi Ajijola, MD, PhD, Principal Investigator — UCLA Health
Locations (1):
- UCLA Health, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Seizure Frequency or Duration Via a Routine Seizure History Used in Clinical Practice.
Time Frame: Following the 4 - week VNS treatment phase to the of the end of study.
Population: Participant only completed first study visit and did not return
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Heart Rate and Blood Pressure in Response to Upright Tilt, Deep Breathing, Valsalva Maneuver and a Cold Pressor Test.
Time Frame: From pre VNS setting changes (baseline) to post VNS setting changes (end of study).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Day
Description: Participant completed only one study visit
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04387435/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04387435/ICF_001.pdf